CLINICAL TRIAL: NCT07297914
Title: Framework for Optimizing, Refining, and Unifying Management of HSCT in Pediatric ALL
Acronym: FORUM2
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORUM2; 2025-522052-13-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-25; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Stem Cell Transplant; Graft -Versus-host-disease
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Graft vs Host Disease | interventions — ruxolitinib; blinatumomab; Cyclophosphamide; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: The FORUM2 study has a flexible design which consists of:
  * Two randomized comparison groups (R1 SUBSTUDY and R2 SUBSTUDY),
  * One stratified cohort (S1 SUBSTUDY),
  * One pilot cohort (P1 SUBSTUDY).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- R1 substudy (Experimental): A phase III, randomized, multi-center study comparing TBI 8 Gy versus TBI 12 Gy in children and young adults with ALL for conditioning of allogeneic HSCT
  Interventions: Radiation: Total Body Irradiation 8 Gy; Radiation: Total Body Irradiation 12 Gy
- R2 substudy (Experimental): A phase III, randomized, open-label multi-center study comparing ruxolitinib plus corticosteroids versus corticosteroids alone in children with ALL and treatment-naïve grade II-IV aGvHD following allogeneic HSCT
  Interventions: Combination Product: Ruxolitinib; Drug: Corticosteroids
- S1 substudy (Experimental): A prospective stratified cohort study comparing between in vivo PT-Cy and ex vivo αβ T-cell depletion in mismatched donor transplantation for pediatric and young adult ALL.
  Interventions: Drug: Cyclophosphamide; Other: αβ T-cells depletion
- P1 substudy (Active Comparator): A phase II, open-label, multi-center study of blinatumomab following allogeneic HSCT for B-lineage ALL in children younger than 2 years not receiving TBI as part of the conditioning regimen
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Radiation: Total Body Irradiation 8 Gy — Total Body Irradiation 8 Gy administered in combination with VP16 as part of the conditioning regimen
  Arms: R1 substudy
Combination Product: Ruxolitinib — Ruxolitinib plus corticosteroids in treatment-naïve acute graft-versus-host disease
  Arms: R2 substudy
Drug: Blinatumomab — Up to four cycles of blinatumomab as post-HSCT maintenance therapy
  Arms: P1 substudy
Drug: Cyclophosphamide — In vivo T-cells depletion/modulation with post-transplant cyclophosphamide
  Arms: S1 substudy
Radiation: Total Body Irradiation 12 Gy — Total Body Irradiation 12 Gy administered in combination with VP16 as part of the conditioning regimen
  Arms: R1 substudy
Drug: Corticosteroids — Corticosteroids alone in treatment-naïve acute graft-versus-host disease
  Arms: R2 substudy
Other: αβ T-cells depletion — Ex vivo graft manipulation based on selective depletion of T-cell receptor αβ (TCR αβ+)/CD19+ lymphocytes from the graft (αβ T-cells depletion)
  Arms: S1 substudy

SUMMARY:
Current therapeutic strategies for high-risk or relapsed ALL patients often involve intensive treatments, including allogeneic hematopoietic stem cell transplantation (HSCT). HSCT remains a cornerstone of therapy, offering curative potential; however, it is associated with considerable risks, including non-relapse mortality (NRM), significant morbidity, and long-term complications that continue to be major concerns.

In response to these challenges, the FORUM consortium has made substantial progress in improving outcomes for children with ALL undergoing HSCT. The consortium focuses on reducing life-threatening and lifelong complications, ultimately aiming to enhance quality of life for these high-risk patients. Building on the robust evidence generated by FORUM1, the FORUM2 study has been designed to further optimize the role of HSCT in ALL across all age groups and donor settings within a harmonized and internationally coordinated framework.

The FORUM2 study introduces a master protocol structure that encompasses multiple hypothesis-driven substudies, each addressing a specific determinant of HSCT outcomes. This design enables simultaneous or sequential evaluation of novel strategies while ensuring uniform governance, endpoint definitions, and data-quality standards. The overarching objective is to refine the role of HSCT in ALL by reducing treatment-related toxicity while preserving the essential graft-versus-leukemia effect.

DETAILED DESCRIPTION:
The key focus areas and objectives include:

* Optimization of conditioning regimens
* Advancements in GvHD prevention and treatment
* Integration of novel immunotherapies
* Improvement of long-term survivorship
* Harmonization of supportive care and post-transplant monitoring
* Expansion of donor availability The FORUM2 study comprises two randomized comparisons (R1 and R2 substudies), one stratified cohort (S1 substudy), and one pilot cohort (P1 substudy). The protocol is structured as a master protocol, with the R1 substudy serving as the central component because it represents the continuation of the FORUM1 study (which compared TBI-based and chemotherapy-based conditioning) and is expected to enroll the majority of patients.

Patients ineligible for the R1 substudy-due to age (<2 years), donor type, physician discretion, or personal preference-will still be included in the master protocol and monitored accordingly. Patients transplanted from a mismatched family donor will be stratified within the S1 substudy. Additionally, patients younger than 2 years of age with B-ALL are eligible for the P1 pilot substudy, which will investigate the use of post-HSCT blinatumomab to reduce relapse incidence in this high-risk population.

Primary and secondary endpoints, general assessment timelines, and supportive care guidelines will remain consistent for both R1 substudy participants and patients included in the broader master protocol. Additional assessments, endpoints, and interventions specific to other study groups are outlined in their respective protocol sections (or appendices) and will be conducted exclusively for patients enrolled in those specific cohorts.

ELIGIBILITY:
Inclusion criteria applicable to all substudies

* Male and female patients with allogenic transplant indication for ALL, as determined by national frontline protocols
* Age ≥3 months to ≤25 years at the time of HSCT.
* Patients must be in complete remission (with <5% blasts and absence of leukemia cells in extramedullary sites) prior to undergoing HSCT.
* Selected donor must be either a matched donor (matched donor category includes 9/10 identical siblings and 10/10 or 9/10 HLA-matched unrelated donors) or a mismatched family donor (≤8/10 HLA match). Either bone marrow or peripheral blood stem cell grafts are permitted. Cord blood is permitted, as well, provided that the unit is at least 6/8 HLA matched and with a cryopreserved cellularity of at least 3x107 nucleated cells/Kg recipient body weight.
* Female patients of childbearing potential must have a negative pregnancy test at screening, and all patients must agree to adhere to effective contraception during the study period.
* Written study informed consent and/or assent from the patient and/or the parent, or guardian

Exclusion criteria applicable to all substudies

* Patients < 3 months and > 25 years of age at the time of HSCT.
* Patients not in complete morphological remission at the time of enrollment.
* Patients with an initial diagnosis of Non-Hodgkin Lymphoma (NHL).
* Patients with ALL as a secondary malignancy.
* Patients with a history of previous autologous or allogeneic HSCT (prior allogeneic transplantation is permitted for subjects receiving post-transplant interventions, such as those enrolled in the R2 and P1 substudies, provided that this is their first allogeneic HSCT).
* Female patients who are pregnant or breast feeding.
* Fertile male or female patients of childbearing potential who do not agree to abstinence or, if sexually active, do not agree to the use of contraception.
* Active clinically uncontrolled bacterial, fungal, parasitic, or viral infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no physical or radiographic signs of infection progression are present.
* Active HBV or HCV infection that requires treatment, or at risk for HBV reactivation (e.g. positive HBsAg). Subjects with negative HbsAg and positive total HB core antibody may be included if HBV DNA is undetectable at the time of screening. Subjects who are positive for HCV antibody are eligible only if polymerase chain reaction test is negative for HCV RNA. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment. Prior serology results are acceptable for determining eligibility.
* Known human immunodeficiency virus infection (HIV).
* Significant respiratory disease including patients who are on mechanical ventilation or who have resting O2 saturation <90% by pulse-oximetry on room-air.
* Presence of severely impaired renal function (confirmed within 72 hours prior to study treatment start) defined by:
* Glomerular Filtration Rate (GFR) < 30 mL/min/1.73 m2 using estimated creatinine clearance calculated by updated bedside Schwartz equation or Cockcroft Gault equation OR
* Renal dialysis requirement
* Clinically significant or uncontrolled cardiac disease including any of the following:
* Uncontrolled hypertension
* New York Heart Association Class III or IV congestive heart failure
* Clinically significant cardiac arrhythmias
* Severe hepatic insufficiency, defined by any of the following:
* Child-Pugh Class C liver disease
* AST (aspartate aminotransferase) or ALT (alanine aminotransferase) levels > 5 times the upper limit of normal (ULN), unless attributable to GvHD
* Total bilirubin > 3.0 mg/dL, unless attributable to GvHD
* INR (International Normalized Ratio) ≥ 1.7
* Clinical evidence of hepatic encephalopathy or ascites
* Presence of severe concomitant constitutional disease that precludes treatment as per protocol, based on the investigator's judgment. Examples include but are not limited to: Down syndrome with severe comorbidities, significant cardiac malformations, and metabolic disorders affecting treatment feasibility.
* Underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would interfere participation in the study, pose a significant risk to the patient or interfere with interpretation of study data.
* Karnofsky or Lansky performance score <50%, indicating significant functional impairment.
* Patients who are unwilling or unable to comply with study procedures, including follow-up requirements and treatment schedules.

Ages: 3 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2032-11-30 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | at year 4
  EFS is defined as the time from randomization (intention-to-treat analysis) or HSCT (per-protocol/as treated) to first failure event defined as follows:
  Failure events are:
  * Relapse
  * Graft failure
  * Death from any cause
  * Diagnosis of a second malignant neoplasm
Overall response rate (ORR) at day 28 | day 28
  Overall response rate (ORR) at day 28 after randomization, defined as the proportion of patients in each arm demonstrating a complete response (CR) or partial response (PR) without requirement for additional systemic therapies for earlier progression, mixed response or nonresponse.
Event Free Survival (EFS) | at year 4
  EFS is defined as the time from HSCT to first failure event defined as follows:
  Failure events are:
  * Relapse
  * Graft failure
  * Death from any cause
  * Diagnosis of a second malignant neoplasm
Cumulative incidence of relapse (CIR) at 2 years after HSCT | 2 years after HSCT
  CIR at 2 years after HSCT in blinatumomab-treated patents and historical controls. CIR is calculated from the time of study enrolment until the date of relapse (defined as either bone marrow aspirate or biopsy with ≥ 5% blasts or as appearance of leukemia cells in an extramedullary site) or last follow-up (death from any cause other than leukemia relapse and secondary malignancies will be considered a competing event)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Locatelli, Professor, Principal Investigator — IRCSS Ospedale Pediatrico Bambino Gesù
Locations (9):
- St'Anna Children Hospital, Vienna, Austria
- University Hospital Motol, Prague, Czechia
- Rigshopsitalet, University Hospital, Copenhagen, Denmark
- HUS-Yhtymae (HUS Helsinki University Hospital), Helsinki, Finland
- Robert- Debré Academic Hospital, Paris, France
- Goethe-Universität, Frankfurt, Germany
- IRCCS Ospedale Pediatrico Bambino Gesù, Roma, RM, Italy
- University Hospital, Oslo, Norway
- University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oostenbrink LVE, Von Asmuth EGJ, Jol-van der Zijde CM, Jansen-Hoogendijk AM, Vervat C, Bredius RGM, Van Tol MJD, Schilham MW, Sedlacek P, Ifversen M, Balduzzi A, Bader P, Peters C, Moes DJAR, Lankester AC. Anti-T-lymphocyte globulin exposure is associated with acute graft-versus-host disease and relapse in pediatric acute lymphoblastic leukemia patients undergoing hematopoietic stem cell transplantation: a multinational prospective study. Haematologica. 2024 Sep 1;109(9):2854-2863. doi: 10.3324/haematol.2023.284632. PMID 38721739
- [Background] Peters C, Dalle JH, Locatelli F, Poetschger U, Sedlacek P, Buechner J, Shaw PJ, Staciuk R, Ifversen M, Pichler H, Vettenranta K, Svec P, Aleinikova O, Stein J, Gungor T, Toporski J, Truong TH, Diaz-de-Heredia C, Bierings M, Ariffin H, Essa M, Burkhardt B, Schultz K, Meisel R, Lankester A, Ansari M, Schrappe M; IBFM Study Group;; von Stackelberg A; IntReALL Study Group; Balduzzi A; I-BFM SCT Study Group; Corbacioglu S; EBMT Paediatric Diseases Working Party; Bader P. Total Body Irradiation or Chemotherapy Conditioning in Childhood ALL: A Multinational, Randomized, Noninferiority Phase III Study. J Clin Oncol. 2021 Feb 1;39(4):295-307. doi: 10.1200/JCO.20.02529. Epub 2020 Dec 17. PMID 33332189
- [Background] Bader P, Potschger U, Dalle JH, Moser LM, Balduzzi A, Ansari M, Buechner J, Gungor T, Ifversen M, Krivan G, Pichler H, Renard M, Staciuk R, Sedlacek P, Stein J, Heusel JR, Truong T, Wachowiak J, Yesilipek A, Locatelli F, Peters C. Low rate of nonrelapse mortality in under-4-year-olds with ALL given chemotherapeutic conditioning for HSCT: a phase 3 FORUM study. Blood Adv. 2024 Jan 23;8(2):416-428. doi: 10.1182/bloodadvances.2023010591. PMID 37738088
- [Background] Kalwak K, Moser LM, Potschger U, Bader P, Kleinschmidt K, Meisel R, Dalle JH, Yesilipek A, Balduzzi A, Krivan G, Goussetis E, Staciuk R, Sedlacek P, Pichler H, Svec P, Gabriel M, Gungor T, Bilic E, Buechner J, Renard M, Vettenranta K, Ifversen M, Diaz-de-Heredia C, Stein J, Toporski J, Bierings M, Peters C, Ansari M, Locatelli F. Comparable outcomes after busulfan- or treosulfan-based conditioning for allo-HSCT in children with ALL: results of FORUM. Blood Adv. 2025 Feb 25;9(4):741-751. doi: 10.1182/bloodadvances.2024014548. PMID 39602342